CLINICAL TRIAL: NCT04648241
Title: A PHASE 3, SINGLE-ARM, OPEN-LABEL STUDY TO EVALUATE THE IMMUNOGENICITY, SAFETY, AND TOLERABILITY OF A TICK-BORNE ENCEPHALITIS VACCINE IN HEALTHY JAPANESE PARTICIPANTS 1 YEAR OF AGE AND OLDER
Brief Title: Study to Evaluate the Immunogenicity, Safety, and Tolerability of a Tick-Borne Encephalitis (TBE) Vaccine in Healthy Japanese Participants 1 Year of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B9371039
Record Dates: First submitted 2020-11-09; First posted 2020-12-01 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Tick-Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ≥16 Years Old (Experimental): TBE vaccine 0.5 mL (intramuscular injection).
  Interventions: Biological: TBE vaccine 0.5 mL
- 1 to <16 Years Old (Experimental): TBE vaccine 0.25ｍL (intramuscular injection).
  Interventions: Biological: TBE vaccine 0.25 mL

INTERVENTIONS:
Biological: TBE vaccine 0.5 mL — TBE vaccine 0.5 mL (intramuscular injection).
  Arms: ≥16 Years Old
Biological: TBE vaccine 0.25 mL — TBE vaccine 0.25 mL (intramuscular injection).
  Arms: 1 to <16 Years Old

SUMMARY:
The main purpose of this study is to provide safety and immunogenicity data in Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female participants ≥1 years old at Visit 1.
* Participants and/or a legally acceptable representative/parent/legal guardian are willing and able to comply with all scheduled visits, vaccination plan, and other study procedures including completion of the e-diary for 7 days for participants after each of 3 vaccinations.
* Participants and/or a legally acceptable representative/parent/legal guardian must be able to be contacted by telephone during study participation.
* Participants and/or a legally acceptable representative/parent/legal guardian are capable of giving signed informed consent.

Exclusion Criteria:

* Major known congenital malformation or serious chronic disorder.
* Known history of TBEV infection.
* Known history of other flavivirus infection (eg, dengue fever, yellow fever, JEV, West Nile virus).
* Known history of infection with HIV, HCV, or HBV.
* Immunocompromised participants with known or suspected immunodeficiency.
* History of autoimmune disease or an active autoimmune disease requiring therapeutic intervention.
* Previous vaccination with any licensed or investigational TBE vaccine, or planned receipt of other flavivirus vaccines apart from JEV vaccine (eg, yellow fever, dengue fever) during the study. Administration of JEV vaccine is prohibited during participation.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Japan (6):
  - Medical Co. LTA PS Clinic, Fukuoka, Fukuoka
  - Azuma kodomo katei clinic, Ebetsu Shi, Hokkaido
  - Watanabe Pediatric Allergy Clinic, Sapporo, Hokkaido
  - Ohigesenseino Kodomo Clinic, Sapporo, Hokkaido
  - SUZURAN Children's Clinic, Sapporo, Hokkaido
  - Childrens clinic of Kose, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Yonekawa M, Watanabe T, Kogawara O, Yoshii C, Yamaji M, Aizawa M, Erber W, Ito S, Jug B, Koelch D, de Solom R, Lockhart SP. Phase 3 immunogenicity and safety study of a tick-borne encephalitis vaccine in healthy Japanese participants 1 year of age and older. Vaccine. 2024 May 10;42(13):3180-3189. doi: 10.1016/j.vaccine.2024.03.071. Epub 2024 Apr 12. PMID 38614954
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9371039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted as part of the Phase 3 clinical development plan to support the use of tick-borne encephalitis (TBE) vaccine 0.5 milliliter (mL) in healthy Japanese adults (greater than or equal to [>=] 16 years old) and 0.25 mL in pediatric participants (>=1 and less than [<] 16 years old) at investigator sites in Japan.
Groups:
- Adults (>=16 Years Old): Participants aged >=16 years old received three doses of 0.5 mL TBE vaccine intramuscularly as Dose 1 on Day 1, Dose 2 between 21 to 35 days after Dose 1 and Dose 3 between 150-365 days after Dose 2. Participants were followed up for safety for 21-35 days after Dose 3.
- Pediatric (1 to <16 Years Old): Participants aged 1 to <16 years old received three doses of 0.25 mL TBE vaccine intramuscularly as Dose 1 on Day 1, Dose 2 between 21 to 35 days after Dose 1 and Dose 3 between 150-365 days after Dose 2. Participants were followed up for safety for 21-35 days after Dose 3.
Period: Overall Study
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Started | 100 | 65
Completed | 99 | 65
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all enrolled participants who received at least 1 dose of the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old) | Total
Number analyzed (Participants) | 100 | 65 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (16.02) | 6.9 (3.89) | 29.5 (22.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 19 | 74
  Male | 45 | 46 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 65 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 100 | 65 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seropositive Participants at 4 Weeks After Dose 3
Description: Seropositivity rate based on the immune response was determined by neutralization test (NT). Participants who achieved tick-borne encephalitis virus (TBEV) NT titers >=1: 10 were considered as seropositive. Exact 2-sided 95% confidence interval (CI) based on the Clopper and Pearson method was presented.
Time Frame: 4 weeks after Dose 3
Population: Evaluable immunogenicity (EI) population: Participants who received all 3 doses of the investigational product, had blood drawn for assay testing within the specified time frame for baseline and 4 weeks after the third vaccination, had valid and determinate assay result (NT titer) at baseline and 4 weeks after the third vaccination visit, were NT seronegative at baseline, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Percentage of participants | 98.0 [92.9 to 99.8] | 100 [94.5 to 100]

2. Primary Outcome: Percentage of Participants With Local Reactions (LR) Within 7 Days After Dose 1
Description: LR:participant or legally acceptable representative/parent/legal guardian using an electronic diary (e-diary). LR included redness, swelling and pain at injection site. Redness and swelling were measured using measuring device units. 1 measuring device unit =0.5 centimeter(cm). Redness and swelling were graded as: for participants >=12 years of age, mild(greater than[>] 2.0 to 5.0 cm), moderate(>5.0 to 10.0 cm) and severe (>10.0 cm); for participants less than (<)12 years of age, mild(>0 to 2.0 cm), moderate(>2.0 to7.0 cm) and severe(>7.0 cm). Pain at the injection site was graded as: for participants >2 years of age, mild(does not interfere with activity), moderate(interferes with activity) and severe(prevents daily activity); for participants less than or equal to (<=)2 years of age, mild(hurts if gently touched) moderate(hurts if gently touched with crying) and severe(causes limitation of limb movement). Exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 7 days after Dose 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants
  Redness: Mild | 2.0 [0.2 to 7.0] | 3.1 [0.4 to 10.7]
  Redness: Moderate | 0 [0.0 to 3.6] | 1.5 [0.0 to 8.3]
  Redness: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Swelling: Mild | 3.0 [0.6 to 8.5] | 3.1 [0.4 to 10.7]
  Swelling: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Swelling: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Pain at the injection site: Mild | 52.0 [41.8 to 62.1] | 36.9 [25.3 to 49.8]
  Pain at the injection site: Moderate | 7.0 [2.9 to 13.9] | 6.2 [1.7 to 15.0]
  Pain at the injection site: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: Local reactions were collected by participant or legally acceptable representative/parent/legal guardian using an e-diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured using measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as: for participants >=12 years of age, mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm); for participants <12 years of age, mild (>0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at the injection site was graded as: for participants >2 years of age, mild (does not interfere with activity), moderate (interferes with activity) and severe (prevents daily activity); for participants <=2 years of age, mild (hurts if gently touched) moderate (hurts if gently touched with crying) and severe (causes limitation of limb movement). Exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 7 days after Dose 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants
  Redness: Mild | 0.0 [0.0 to 3.6] | 3.1 [0.4 to 10.7]
  Redness: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Redness: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Swelling: Mild | 0 [0.0 to 3.6] | 1.5 [0.0 to 8.3]
  Swelling: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Swelling: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]
  Pain at the injection site: Mild | 40.0 [30.3 to 50.3] | 24.6 [14.8 to 36.9]
  Pain at the injection site: Moderate | 4.0 [1.1 to 9.9] | 1.5 [0.0 to 8.3]
  Pain at the injection site: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 5.5]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: as for outcome 3
Time Frame: Within 7 days after Dose 3
Population: Safety analysis population included all enrolled participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Percentage of participants
  Redness: Mild | 2.0 [0.2 to 7.1] | 7.7 [2.5 to 17.0]
  Redness: Moderate | 0 [0.0 to 3.7] | 0 [0.0 to 5.5]
  Redness: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 5.5]
  Swelling: Mild | 1.0 [0.0 to 5.5] | 6.2 [1.7 to 15.0]
  Swelling: Moderate | 1.0 [0.0 to 5.5] | 3.1 [0.4 to 10.7]
  Swelling: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 5.5]
  Pain at the injection site: Mild | 33.3 [24.2 to 43.5] | 30.8 [19.9 to 43.4]
  Pain at the injection site: Moderate | 3.0 [0.6 to 8.6] | 4.6 [1.0 to 12.9]
  Pain at the injection site: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 5.5]

5. Primary Outcome: Percentage of Participants With Systemic Events (SE) Within 7 Days After Dose 1
Description: SE:participants or legally acceptable representative/parent/legal guardian using e-diary & included fever:temperature >=37.5 degree Celsius(C)&categorized as 37.5to38.4, 38.5 to 38.9,39.0 to 40.0,>40.0 degree C.Fatigue, headache, muscle pain, joint pain: mild(didn't interfere with activity), moderate(some interference with activity), severe(prevented daily activity). Vomiting: mild(1-2 times in 24 hours[hrs]), moderate(>2 times in 24hrs), severe(required intravenous hydration). Diarrhea: mild(2-3 loose stools in 24hrs), moderate(4-5 loose stools in 24hrs), severe(6 or more loose stools in 24hrs). Decreased appetite:mild(decreased interest in eating),moderate(decreased oral intake), severe(refusal to feed).Drowsiness: mild(Increased sleeping bouts),moderate(slightly subdued interfering with daily activity),severe(disabling not interested in usual daily activity).Irritability:mild(easily consolable), moderate(required increased attention),severe(inconsolable, crying can't be comforted).
Time Frame: Within 7 days after Dose 1
Population: Safety analysis population included all enrolled participants who received at least 1 dose of the investigational product. Here, 'Number Analyzed' signifies those participants who were evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pediatric (3 to 15 Years Old): Participants aged 1 to <16 years old received three doses of 0.25 mL TBE vaccine intramuscularly as Dose 1 on Day 1, Dose 2 between 21 to 35 days after Dose 1 and Dose 3 between 150-365 days after Dose 2. Participants were followed up for safety for 21-35 days after Dose 3.
- Pediatric (1 to 2 Years Old): Participants aged 1 to 2 years old received three doses of 0.25 mL TBE vaccine intramuscularly as Dose 1 on Day 1, Dose 2 between 21 to 35 days after Dose 1 and Dose 3 between 150-365 days after Dose 2. Participants were followed up for safety for 21-35 days after Dose 3.
Arm/Group | Adults (>=16 Years Old) | Pediatric (3 to 15 Years Old) | Pediatric (1 to 2 Years Old)
Number analyzed (Participants) | 100 | 57 | 8
Percentage of participants
  Fever: >=37.5 degree C | 2.0 [0.2 to 7.0] | 5.3 [1.1 to 14.6] | 25.0 [3.2 to 65.1]
  Fever: 37.5 to 38.4 degree C | 2.0 [0.2 to 7.0] | 3.5 [0.4 to 12.1] | 25.0 [3.2 to 65.1]
  Fever: 38.5 to 38.9 degree C | 0 [0.0 to 3.6] | 1.8 [0.0 to 9.4] | 0 [0.0 to 36.9]
  Fever: 39.0 to 40.0 degree C | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fever: >40.0 degree C | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fatigue: Mild: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Mild | 11.0 [5.6 to 18.8] | 8.8 [2.9 to 19.3] |
  Fatigue: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Moderate | 5.0 [1.6 to 11.3] | 1.8 [0.0 to 9.4] |
  Fatigue: Severe: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Headache: Mild: number analyzed (Participants) | 100 | 57 | 0
  Headache: Mild | 7.0 [2.9 to 13.9] | 7.0 [1.9 to 17.0] |
  Headache: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Headache: Moderate | 6.0 [2.2 to 12.6] | 1.8 [0.0 to 9.4] |
  Headache: Severe: number analyzed (Participants) | 100 | 57 | 0
  Headache: Severe | 0 [0.0 to 3.6] | 1.8 [0.0 to 9.4] |
  Vomiting: Mild: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Mild | 1.0 [0.0 to 5.4] | 0 [0.0 to 6.3] |
  Vomiting: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Moderate | 1.0 [0.0 to 5.4] | 0 [0.0 to 6.3] |
  Vomiting: Severe: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Diarrhea: Mild: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Mild | 7.0 [2.9 to 13.9] | 8.8 [1.9 to 19.3] |
  Diarrhea: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Moderate | 2.0 [0.2 to 7.0] | 0 [0.0 to 6.3] |
  Diarrhea: Severe: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Muscle pain: Mild: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Mild | 16.0 [9.4 to 24.7] | 5.3 [1.1 to 14.6] |
  Muscle pain: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Moderate | 3.0 [0.6 to 8.5] | 0 [0.0 to 6.3] |
  Muscle pain: Severe: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Joint pain: Mild: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Mild | 4.0 [1.1 to 9.9] | 0 [0.0 to 6.3] |
  Joint pain: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Moderate | 3.0 [0.6 to 8.5] | 0 [0.0 to 6.3] |
  Joint pain: Severe: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Decreased appetite: Mild: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Mild |  |  | 0 [0.0 to 36.9]
  Decreased appetite: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Moderate |  |  | 12.5 [0.3 to 52.7]
  Decreased appetite: Severe: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Severe |  |  | 0 [0.0 to 36.9]
  Drowsiness: Mild: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Mild |  |  | 25.0 [3.2 to 65.1]
  Drowsiness: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Moderate |  |  | 0 [0.0 to 36.9]
  Drowsiness: Severe: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Severe |  |  | 0 [0.0 to 36.9]
  Irritability: Mild: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Mild |  |  | 12.5 [0.3 to 52.7]
  Irritability: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Moderate |  |  | 12.5 [0.3 to 52.7]
  Irritability: Severe: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Severe |  |  | 0 [0.0 to 36.9]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: SE:participants or a legally acceptable representative/parent/legal guardian using e-diary and included fever:temperature >=37.5 degreeC & categorized as 37.5 to 38.4,38.5 to 38.9,39.0 to 40.0,>40.0 degreeC.Fatigue, headache, muscle pain, joint pain: mild(didn't interfere with activity),moderate(some interference with activity), severe(prevented daily activity). Vomiting: mild(1-2 times in 24 hours[hrs]), moderate(>2 times in 24hrs),severe(required intravenous hydration).Diarrhea: mild(2-3 loose stools in 24hrs), moderate(4-5 loose stools in 24hrs), severe(6 or more loose stools in 24hrs). Decreased appetite: mild(decreased interest in eating), moderate(decreased oral intake), severe(refusal to feed). Drowsiness: mild(Increased sleeping bouts), moderate(slightly subdued interfering with daily activity), severe(disabling not interested in usual daily activity).Irritability: mild(easily consolable), moderate(required increased attention),severe(inconsolable, crying can't be comforted).
Time Frame: Within 7 days after Dose 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pediatric (1 to 2 Years Old): Participants received three doses of 0.25 mL TBE vaccine intramuscularly as Dose 1 on Day 1, Dose 2 between 21 to 35 days after Dose 1 and Dose 3 between 150-365 days after Dose 2. Participants were followed up for safety for 21-35 days after Dose 3.
Arm/Group | Adults (>=16 Years Old) | Pediatric (3 to 15 Years Old) | Pediatric (1 to 2 Years Old)
Number analyzed (Participants) | 100 | 57 | 8
Percentage of participants
  Fever: >=37.5 degree C | 1.0 [0.0 to 5.4] | 7.0 [1.9 to 17.0] | 0 [0.0 to 36.9]
  Fever: 37.5 to 38.4 degree C | 1.0 [0.0 to 5.4] | 3.5 [0.4 to 12.1] | 0 [0.0 to 36.9]
  Fever: 38.5 to 38.9 degree C | 0 [0.0 to 3.6] | 3.5 [0.4 to 12.1] | 0 [0.0 to 36.9]
  Fever: 39.0 to 40.0 degree C | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fever: >40.0 degree C | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fatigue: Mild: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Mild | 7.0 [2.9 to 13.9] | 1.8 [0.0 to 9.4] |
  Fatigue: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Moderate | 1.0 [0.0 to 5.4] | 0 [0.0 to 6.3] |
  Fatigue: Severe: number analyzed (Participants) | 100 | 57 | 0
  Fatigue: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Headache: Mild: number analyzed (Participants) | 100 | 57 | 0
  Headache: Mild | 10.0 [4.9 to 17.6] | 0 [0.0 to 6.3] |
  Headache: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Headache: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Headache: Severe: number analyzed (Participants) | 100 | 57 | 0
  Headache: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Vomiting: Mild: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Mild | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Vomiting: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Vomiting: Severe: number analyzed (Participants) | 100 | 57 | 0
  Vomiting: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Diarrhea: Mild: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Mild | 4.0 [1.1 to 9.9] | 7.0 [1.9 to 17.0] |
  Diarrhea: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Moderate | 1.0 [0.0 to 5.4] | 0 [0.0 to 6.3] |
  Diarrhea: Severe: number analyzed (Participants) | 100 | 57 | 0
  Diarrhea: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Muscle pain: Mild: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Mild | 2.0 [0.2 to 7.0] | 1.8 [0.0 to 9.4] |
  Muscle pain: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Muscle pain: Severe: number analyzed (Participants) | 100 | 57 | 0
  Muscle pain: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Joint pain: Mild: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Mild | 1.0 [0.0 to 5.4] | 0 [0.0 to 6.3] |
  Joint pain: Moderate: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Moderate | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Joint pain: Severe: number analyzed (Participants) | 100 | 57 | 0
  Joint pain: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 6.3] |
  Decreased appetite: Mild: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Mild |  |  | 0 [0.0 to 36.9]
  Decreased appetite: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Moderate |  |  | 0 [0.0 to 36.9]
  Decreased appetite: Severe: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Severe |  |  | 0 [0.0 to 36.9]
  Drowsiness: Mild: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Mild |  |  | 12.5 [0.3 to 52.7]
  Drowsiness: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Moderate |  |  | 0 [0.0 to 36.9]
  Drowsiness: Severe: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Severe |  |  | 0 [0.0 to 36.9]
  Irritability: Mild: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Mild |  |  | 0 [0.0 to 36.9]
  Irritability: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Moderate |  |  | 0 [0.0 to 36.9]
  Irritability: Severe: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Severe |  |  | 0 [0.0 to 36.9]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: Systemic events collected by participant using e-diary and included fever defined as temperature >=37.5 degree C and categorized as 37.5 to 38.4, 38.5 to 38.9, 39.0 to 40.0, >40.0 degree C. Fatigue, headache, muscle pain, joint pain: mild(didn't interfere with activity), moderate(some interference with activity), severe(prevented daily activity). Vomiting: mild(1-2 times in 24 hours[hrs]), moderate(>2 times in 24hrs), severe(required intravenous hydration). Diarrhea: mild(2-3 loose stools in 24hrs), moderate(4-5 loose stools in 24hrs), severe(6 or more loose stools in 24hrs). Decreased appetite: mild(decreased interest in eating), moderate(decreased oral intake), severe(refusal to feed). Drowsiness: mild(Increased sleeping bouts), moderate(slightly subdued interfering with daily activity), severe(disabling not interested in usual daily activity). Irritability: mild(easily consolable), moderate(required increased attention), severe(inconsolable, crying can't be comforted).
Time Frame: Within 7 days after Dose 3
Population: Safety analysis population included all enrolled participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and 'Number Analyzed' signifies those participants who were evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (3 to 15 Years Old) | Pediatric (1 to 2 Years Old)
Number analyzed (Participants) | 99 | 57 | 8
Percentage of participants
  Fever: >=37.5 degree C | 1.0 [0.0 to 5.5] | 10.5 [4.0 to 21.5] | 12.5 [0.3 to 52.7]
  Fever: 37.5 to 38.4 degree C | 0 [0.0 to 3.7] | 8.8 [2.9 to 19.3] | 12.5 [0.3 to 52.7]
  Fever: 38.5 to 38.9 degree C | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fever: 39.0 to 40.0 degree C | 0 [0.0 to 3.7] | 1.8 [0.0 to 9.4] | 0 [0.0 to 36.9]
  Fever: >40.0 degree C | 0 [0.0 to 3.7] | 0 [0.0 to 6.3] | 0 [0.0 to 36.9]
  Fatigue: Mild: number analyzed (Participants) | 99 | 57 | 0
  Fatigue: Mild | 9.1 [4.2 to 16.6] | 1.8 [0.0 to 9.4] |
  Fatigue: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Fatigue: Moderate | 2.0 [0.2 to 7.1] | 5.3 [1.1 to 14.6] |
  Fatigue: Severe: number analyzed (Participants) | 99 | 57 | 0
  Fatigue: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 6.3] |
  Headache: Mild: number analyzed (Participants) | 99 | 57 | 0
  Headache: Mild | 9.1 [4.2 to 16.6] | 5.3 [1.1 to 14.6] |
  Headache: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Headache: Moderate | 1.0 [0.0 to 5.5] | 3.5 [0.4 to 12.1] |
  Headache: Severe: number analyzed (Participants) | 99 | 57 | 0
  Headache: Severe | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] |
  Vomiting: Mild: number analyzed (Participants) | 99 | 57 | 0
  Vomiting: Mild | 2.0 [0.2 to 7.1] | 1.8 [0.0 to 9.4] |
  Vomiting: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Vomiting: Moderate | 0 [0.0 to 3.7] | 1.8 [0.0 to 9.4] |
  Vomiting: Severe: number analyzed (Participants) | 99 | 57 | 0
  Vomiting: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 6.3] |
  Diarrhea: Mild: number analyzed (Participants) | 99 | 57 | 0
  Diarrhea: Mild | 5.1 [1.7 to 11.4] | 5.3 [1.1 to 14.6] |
  Diarrhea: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Diarrhea: Moderate | 0 [0.0 to 3.7] | 3.5 [0.4 to 12.1] |
  Diarrhea: Severe: number analyzed (Participants) | 99 | 57 | 0
  Diarrhea: Severe | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] |
  Muscle pain: Mild: number analyzed (Participants) | 99 | 57 | 0
  Muscle pain: Mild | 3.0 [0.6 to 8.6] | 1.8 [0.0 to 9.4] |
  Muscle pain: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Muscle pain: Moderate | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] |
  Muscle pain: Severe: number analyzed (Participants) | 99 | 57 | 0
  Muscle pain: Severe | 0 [0.0 to 3.7] | 0 [0.0 to 6.3] |
  Joint pain: Mild: number analyzed (Participants) | 99 | 57 | 0
  Joint pain: Mild | 0 [0.0 to 3.7] | 5.3 [1.1 to 14.6] |
  Joint pain: Moderate: number analyzed (Participants) | 99 | 57 | 0
  Joint pain: Moderate | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] |
  Joint pain: Severe: number analyzed (Participants) | 99 | 57 | 0
  Joint pain: Severe | 1.0 [0.0 to 5.5] | 0 [0.0 to 6.3] |
  Decreased appetite: Mild: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Mild |  |  | 12.5 [0.3 to 52.7]
  Decreased appetite: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Moderate |  |  | 0 [0.0 to 36.9]
  Decreased appetite: Severe: number analyzed (Participants) | 0 | 0 | 8
  Decreased appetite: Severe |  |  | 0 [0.0 to 36.9]
  Drowsiness: Mild: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Mild |  |  | 25.0 [3.2 to 65.1]
  Drowsiness: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Moderate |  |  | 0 [0.0 to 36.9]
  Drowsiness: Severe: number analyzed (Participants) | 0 | 0 | 8
  Drowsiness: Severe |  |  | 0 [0.0 to 36.9]
  Irritability: Mild: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Mild |  |  | 0 [0.0 to 36.9]
  Irritability: Moderate: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Moderate |  |  | 0 [0.0 to 36.9]
  Irritability: Severe: number analyzed (Participants) | 0 | 0 | 8
  Irritability: Severe |  |  | 0 [0.0 to 36.9]

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Dose 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention. Exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 1 month after Dose 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants | 6.0 [2.2 to 12.6] | 21.5 [12.3 to 33.5]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Dose 2
Description: as for outcome 8
Time Frame: Within 1 month after Dose 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants | 2.0 [0.2 to 7.0] | 10.8 [4.4 to 20.9]

10. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Dose 3
Description: as for outcome 8
Time Frame: Within 1 month after Dose 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Percentage of participants | 6.1 [2.3 to 12.7] | 29.2 [18.6 to 41.8]

11. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Any Dose
Description: as for outcome 8
Time Frame: Within 1 month after any Dose
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants | 14.0 [7.9 to 22.4] | 41.5 [29.4 to 54.4]

12. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Throughout the Study
Description: An SAE was defined as any untoward medical occurrence that, at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect or that is considered to be an important medical event. Percentage of participants with SAEs and the exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: From Day 1 up to end of study (up to approximately 13 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants | 2.0 [0.2 to 7.0] | 1.5 [0.0 to 8.3]

13. Secondary Outcome: Percentage of Seropositive Participants at 4 Weeks After Dose 2
Description: Seropositivity rate based on the immune response was determined by NT. Participants who achieved TBEV NT titers >=1: 10 were considered as seropositive. Exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: 4 weeks after Dose 2
Population: Evaluable immunogenicity (EI) population for the second dose: Participants who received the first 2 doses of the investigational product, had blood drawn for assay testing within the specified time frame for baseline and 4 weeks after the second vaccination, had valid and determinate assay result (NT titer) at baseline and 4 weeks after the second vaccination visit, were NT seronegative at baseline, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Percentage of participants | 93 [86.1 to 97.1] | 92.3 [83.0 to 97.5]

14. Secondary Outcome: Geometric Mean Titers (GMTs) of TBEV Neutralizing Antibody Titers at 4 Weeks After Dose 2 and Dose 3
Description: GMTs and associated 2-sided 95% CIs were calculated as the mean of the assay results on the natural logarithmic scale based on Student's t distribution and then exponentiating the results. The lower limit of quantitation (LLOQ) value for NT was 5. Assay results below the LLOQ were set to 0.5 × LLOQ.
Time Frame: 4 weeks after Dose 2 and Dose 3
Population: EI population: Participants who received all 3 doses of the investigational product, had blood drawn for assay testing within specified time frame for baseline and 4 weeks after the third vaccination, had valid and determinate assay result (NT titer) at baseline and 4 weeks after the third vaccination visit, were NT seronegative at baseline, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Titer
  4 Weeks after Dose 2 | 28.2 [23.5 to 33.8] | 29.4 [23.3 to 37.0]
  4 Weeks after Dose 3 | 80.1 [65.1 to 98.5] | 233.1 [187.9 to 289.1]

15. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of TBEV Neutralizing Antibody Titers at 4 Weeks After Dose 2 as Compared to Baseline
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). The LLOQ value for NT was 5. Assay results below the LLOQ were set to 0.5 × LLOQ.
Time Frame: From Baseline to 4 weeks after Dose 2
Population: Evaluable immunogenicity population for the second dose: Participants who received the first 2 doses of the investigational product, had blood drawn for assay testing within the specified time frame for baseline and 4 weeks after the second vaccination, had valid and determinate assay result (NT titer) at baseline and 4 weeks after the second vaccination visit, were NT seronegative at baseline, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 100 | 65
Fold rise | 11.2 [9.3 to 13.4] | 11.8 [9.3 to 14.8]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of TBEV Neutralizing Antibody Titers at 4 Weeks After Dose 3 as Compared to Baseline
Description: as for outcome 15
Time Frame: From Baseline to 4 weeks after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Fold rise | 32.0 [26.0 to 39.4] | 93.2 [75.2 to 115.6]

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of TBEV Neutralizing Antibody Titers at 4 Weeks After Dose 3 as Compared to 4 Weeks After Dose 2
Description: as for outcome 15
Time Frame: From 4 weeks after Dose 2 to 4 weeks after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Fold rise | 2.8 [2.3 to 3.5] | 7.9 [6.2 to 10.2]

18. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers >= Lower Limit of Quantification (LLOQ)
Description: The LLOQ value for NT was 5. Assay results below the LLOQ were set to 0.5 × LLOQ. Percentage of participants with NT>=LLOQ and exact 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Before Dose 1, 4 weeks after Dose 2, Before Dose 3 and 4 weeks after Dose 3
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
Number analyzed (Participants) | 99 | 65
Percentage of Participants
  Before Dose 1 | 0 [0.0 to 3.7] | 0 [0.0 to 5.5]
  4 Weeks after Dose 2 | 96.0 [90.0 to 98.9] | 98.5 [91.7 to 100.0]
  Before Dose 3 | 63.6 [53.4 to 73.1] | 86.2 [75.3 to 93.5]
  4 Weeks after Dose 3 | 99.0 [94.5 to 100.0] | 100.0 [94.5 to 100.0]

ADVERSE EVENTS:
Time Frame: All-Cause mortality and SAEs: from Day 1 up to end of study (up to approximately 13 months); Other AEs (non-systematic assessment): up to 1 month after each Dose; Local reactions and systemic events (systematic assessment, included in other AEs): within 7 days after each Dose
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis population included all enrolled participants who received at least 1 dose of the investigational product.
Arm/Group | Adults (>=16 Years Old) | Pediatric (1 to <16 Years Old)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/65
Serious Adverse Events (participants affected / at risk) | 2/100 | 1/65
Other Adverse Events (participants affected / at risk) | 76/100 | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (>=16 Years Old) (N=100) | Pediatric (1 to <16 Years Old) (N=65)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (>=16 Years Old) (N=100) | Pediatric (1 to <16 Years Old) (N=65)
Blepharitis (Eye disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 15 | 12
Vomiting (VOMITING) (Gastrointestinal disorders) | 4 | 2
Fatigue (FATIGUE) (General disorders) | 27 | 9
Injection site erythema (REDNESS) (General disorders) | 3 | 7
Injection site pain (PAIN) (General disorders) | 68 | 43
Injection site swelling (SWELLING) (General disorders) | 4 | 9
Pyrexia (FEVER) (General disorders) | 3 | 13
Vessel puncture site bruise (General disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 3
Empyema (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 11
Otitis externa (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 1 | 8
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 10 | 3
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 22 | 4
Headache (HEADACHE) (Nervous system disorders) | 23 | 9
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 0 | 3
Irritability (IRRITABILITY) (Psychiatric disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT04648241/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT04648241/SAP_001.pdf